CLINICAL TRIAL: NCT01155986
Title: Lidocaine 5% Medicated Plaster for the Topical Treatment of Localized Chronic Postoperative Neuropathic Pain.
Brief Title: Lidocaine 5% Medicated Plaster in Chronic Neuropathic Postoperative Pain
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial was stopped due to difficult enrolment
Sponsor: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 761541; 2009-016337-10 (EudraCT Number)
Record Dates: First submitted 2010-07-01; First posted 2010-07-02 (Estimated); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Pain; Chronic Pain; Neuropathic Pain; Postoperative Pain
Keywords: analgesic; analgesics; pain; chronic pain; localized pain; focal pain; neuropathic pain; postoperative pain; topical analgesia
MeSH Terms: conditions — Pain; Chronic Pain; Neuralgia; Pain, Postoperative | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo Plaster (Placebo Comparator): Active Comparator
  Interventions: Drug: Placebo topical plaster
- Lidocaine Plaster (Active Comparator)
  Interventions: Drug: Lidocaine 5% medicated plaster

INTERVENTIONS:
Drug: Lidocaine 5% medicated plaster — Topical hydrogel plaster (700mg lidocaine)
  Other Names: Versatis(R)
  Arms: Lidocaine Plaster
Drug: Placebo topical plaster — Topical hydrogel plaster
  Arms: Placebo Plaster

SUMMARY:
The purpose of this trial is to investigate the efficacy and safety of lidocaine 5% medicated plaster in localized chronic post-operative neuropathic pain in comparison to placebo plaster.

DETAILED DESCRIPTION:
Some patients who undergo different types of surgery develop distressing and long-lasting pain. This pain is often characterized by signs such as: allodynia (a pain due to a stimulus which does not normally provoke pain), dysesthesia (unpleasant, abnormal sense of touch). Patients describe symptoms of burning or electrical type sensation. In some cases this type of chronic pain can still be present after 3 months or more following surgery.This clinical trial will assess the efficacy and safety profile of lidocaine 5% medicated plaster in comparison to placebo plaster in patients.

This trial is a randomized, double-blind (neither investigator nor patient will know which treatment was received), placebo-controlled, parallel-group, multicenter trial to evaluate topical analgesic treatment of chronic neuropathic pain after surgery. The trial will include a screening phase and a treatment phase, during which subjects will be treated with either 5% lidocaine medicated plaster, or a placebo plaster pain intensity will be assessed on a daily basis. Subsequently there will be a follow-up phase. Pain intensity numeric rating scale (PI) will be collected via the numeric rating scale and averaged. Safety evaluations include monitoring of adverse events, physical examinations, and clinical laboratory tests.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects with >= 18 years of age
* Intact skin in the area of topical treatment
* Patients suffering from moderate to severe ( 5 or more points on an 11 point Numerical Rating Scale where 10 is the worst possible pain, and 0 indicates no pain) chronic daily postoperative neuropathic pain for the past 6 to 24 months.
* Patients should have symptoms for example allodynia (a pain due to a stimulus which does not normally provoke pain); and or dysesthesia (unpleasant, abnormal sense of touch).

Exclusion Criteria:

* Contraindications to lidocaine 5% medicated plaster, or paracetamol
* Evidence or history of alcohol, medication or drug abuse and/or dependency in the past 3 years.
* Evidence or history (during the past 3 years) of epilepsy, neurotic personality, psychiatric illness, or suicide risk.
* Pregnant or breastfeeding women
* Women of childbearing potential who are sexually active without satisfactory contraception for at least 28 days prior to enrollment, during the trial, and until 28 days after the follow-up visit.
* Severe renal, hepatic or heart disorder.
* Surgery in the past 3 months before screening.
* Anticipated need for surgery during the trial, requiring at least regional or general anesthesia.
* Pending litigation due to chronic pain or disability.
* Participation in another trial of investigational medicinal products or devices parallel to or less than 1 month before entry into the trial, or previous participation in this trial.
* Presence of other severe pain that could confound the assessment or self- evaluation of the localized postoperative neuropathic pain.
* For patients with chronic postoperative neuropathic pain related to a surgery due to tumors: suspected residual tumor or metastases, chemotherapy or radiotherapy for treatment of tumor(s).
* Total anesthesia in the area of localized chronic pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2010-08; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Analgesic efficacy of lidocaine 5% medicated plaster in comparison to placebo in subjects with moderate to severe localized chronic postoperative neuropathic pain | daily assessments over 4 weeks
  Participants will be selected based on their medical history and clinical examination. A questionnaire called DN4, which stands for 'douleur neuropathique 4' (i.e., '4 questions neuropathic pain will be used to identify subjects with neuropathic pain.) Pain will be assessed on and 11-point numerical rating scale (0 = no pain, 10 = worst pain imaginable).
  Efficacy of the treatment (i.e., reduction of neuropathic pain) will be evaluated with the 11-point numeric rating scale (NRS).

SECONDARY OUTCOMES:
Effect of lidocaine 5% medicated plaster on quality of life | 4 weeks
  EuroQol-5 Dimension Scores
Neuropathic Pain Symptoms | 4 weeks
  Changes in severity of various neuropathic pain symptoms, e.g. allodynia, will be recorded by the Neuropathic Pain Symptom Inventory (NPSI) and neurological examinations
Incidence of adverse events | up to 44 days
  Measurement of adverse events including those derived from laboratory data or vital signs measurements.
Hospital Anxiety and Depression Scale | 4 weeks
Subject's Global Impression of Change | 4 weeks
Treatment Satisfaction Questionnaire for Medication | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jean Bruxelle, Principal Investigator — Fondation Ophtalmologique Adolphe de Rotschild, Service de Neurochirurgie, CEntre d'Evaluation et de Traitement de la Douleur
Locations (22):
- France (22):
  - Site 31, Abbeville
  - Site 26, Bayonne
  - Site 34, Bobigny
  - Site 35, Bordeaux
  - Site 12, Boulogne-Billancourt
  - Site 24, Brest
  - Site 15, Châteauroux
  - Site 30, Corbeil-Essonnes
  - Site 39, La Roche-sur-Yon
  - Site 23, Lille
  - Site 17, Limoges
  - Site 21, Marseille
  - Site 33, Montauban
  - Site 14, Nice
  - Site 18, Orléans
  - Site 27, Paris
  - Site 36, Paris
  - Site 22, Rennes
  - Site 20, Saint-Etienne
  - Site 19, Saint-Genis-Laval
  - Site 38, Tours
  - Site 28, Voiron